CLINICAL TRIAL: NCT02860481
Title: FSH-R (Follicle-stimulating Hormone Receptor ): Diagnostic Application for Localized Tumors in Cancerology
Brief Title: FSH-R : Diagnostic Application for Localized Tumors in Cancerology
Acronym: FRACTal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IC 2012-09
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2016-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- first cohort : first 100 patients (Other): first cohort : first 100 patients 10 patients with ovarian and/or endometrial cancer 10 patients with colorectal cancer 10 patients with head and neck cancer 10 patients with uveal melanoma 40 patients with invasive breast cancer 10 patients with breast ductal carcinoma in situ 10 patients with other tumor type
  Interventions: Procedure: blood sample for FSHR analysis
- second cohort : 100 patients (Other): Patients with breast cancer of with ovarian and/or endometrial cancer
  Interventions: Procedure: blood sample for FSHR analysis

INTERVENTIONS:
Procedure: blood sample for FSHR analysis
  Arms: first cohort : first 100 patients
Procedure: blood sample for FSHR analysis
  Arms: second cohort : 100 patients

SUMMARY:
FRACTal study is the first exploration of detection of FSHR as a blood biomarker for the diagnosis of cancer.

A first cohort will explore several common (e.g. breast, prostate) or rare (e.g. uveal melanoma) cancers, that are frequently treated at Institut Curie. This first cohort will include n=10 patients per histological type except for breast cancer (n=50). 100 patients are expected in this cohort.

A second cohort will explore the more promising histological type (if any) in term of incidence of detection. 100 patients are expected for this second cohort.

ELIGIBILITY:
Inclusion criteria

1. Patient diagnosed with localized cancer and corresponding to the different types explored. The cancer can be already diagnosed or not (strong suspicion)
2. Age> 18
3. Written informed consent

Exclusion criteria

1. Previous treatment for the tumoral disease
2. Personal history of cancer diagnosis in the last 10 years
3. Pregnant and/or breastfeeding women
4. Person deprived of liberty or under guardianship (including curatorship)
5. psychiatric illness/social situation that would interfere with the protocol or limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-11; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
sensitivity of blood FSH R detection in cancer patients | end of the study, up to two years

SECONDARY OUTCOMES:
variability of blood FSH-R in the same tumoral type and between different tumoral types | end of the study, up to two years
comparison of blood FSH-R with blood from healthy donor | end of the study, up to two years

CONTACTS AND LOCATIONS:
Overall Officials: François Clément Bidard, MD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Centre René Huguenin, Saint-Cloud

IPD SHARING:
Plan to Share IPD: No